CLINICAL TRIAL: NCT03919175
Title: A Phase 2 Study of Umbralisib and Rituximab as Initial Therapy for Patients With Follicular Lymphoma and Marginal Zone Lymphoma
Brief Title: Umbralisib and Rituximab as Initial Therapy for Patients With Follicular Lymphoma and Marginal Zone Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Umbralisib development terminated; closed to accrual 8/29/2022
Sponsor: Massachusetts General Hospital (Other)
Collaborators: TG Therapeutics (Unknown)
Responsible Party: Principal Investigator, Jacob Soumerai, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-011
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma; Follicular Lymphoma; Follicular Lymphoma, Grade 1; Follicular Lymphoma Grade 2; Follicular Lymphoma Grade IIIa; Marginal Zone Lymphoma; Marginal Zone B Cell Lymphoma
Keywords: Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — umbralisib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Umbralisib+Rituximab (Experimental): * A treatment cycle is defined as 28 consecutive days.
  * Umbralisib will be administered at 800 mg by mouth once daily on days 1-28 of cycles 1-24.
  * Rituximab will be administered at 375 mg/m2 by intravenous infusion on Cycle 1 Day 1 and may be administered at 375 mg/m2 by intravenous infusion or at 1400 mg by subcutaneous injection on days 8, 15, 22 of cycle 1, day 1 of cycles 2 to 6, then every 8 weeks starting on day 1 of cycle 7 until completion of 24 cycles of umbralisib (i.e. every other cycle for 18 cycles or 9 doses, for a total of 15 doses of rituximab), or until progression or intolerance.
  Interventions: Drug: Umbralisib; Drug: Rituximab

INTERVENTIONS:
Drug: Umbralisib — Umbralisib is an investigational drug which blocks a protein called PI3K. PI3K is a protein that plays a role in the way cells grow. In this type of cancer, PI3K is increased and more active than usual. This helps the cancer cells to grow and survive.
  Other Names: TGR-1202
Drug: Rituximab — Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells
  Other Names: MabThera

SUMMARY:
This research is being done to assess Umbralisib and Rituximab as a first line therapy for Follicular Lymphoma or Marginal Zone Lymphoma.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved Umbralisib as a treatment for any disease.

The FDA has approved Rituximab as a treatment option for this disease.

Umbralisib is an investigational drug which blocks a protein called PI3K. PI3K is a protein that plays a role in the way cells grow. In this type of cancer, PI3K is increased and more active than usual. This helps the cancer cells to grow and survive. Early clinical trials have shown that Umbralisib can kill cancer cells in some patients and cause their tumors to shrink.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed follicular lymphoma grade 1-3A or marginal zone lymphoma by WHO criteria.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter [LDi] to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥15 mm in LDi for nodal disease or >10 mm in LDi for extranodal lesions.
* Requires therapy based on: symptomatic disease, threatened end-organ dysfunction, compressive disease, cytopenias secondary to lymphoma, bulky disease (defined as any site ≥7 cm, or 3 or more sites ≥3cm), or steady progression.
* For patients with follicular lymphoma: No prior systemic therapy for follicular lymphoma. Prior radiation to a single site of disease is allowed if completed at least 2 weeks prior to initiation of protocol therapy and there are additional sites of measurable disease outside of the radiation field.
* For patients with marginal zone lymphoma: No prior systemic therapy for marginal zone lymphoma. Prior radiation or surgical resection is allowed if there are additional sites of measurable disease outside of the radiation field. Prior radiation must be completed at least 2 weeks prior to initiation of protocol therapy. Prior H. pylori eradication therapy is allowed.
* Age >18 years.
* ECOG performance status ≤2
* Participants must have adequate organ function as defined below:

  * total bilirubin <1.5 x institutional upper limit of normal (ULN) or <3 x ULN if considered due to Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥30 mL/min for participants with creatinine levels above institutional normal.
* Participants must have adequate marrow function as defined below (unless abnormalities are considered related to marrow involvement by lymphoma):

  * absolute neutrophil count ≥1,000/mcL (500/mcL is acceptable if due to marrow involvement by lymphoma)
  * platelets ≥70,000/mcL(30,000/mcL is acceptable if due to marrow involvement by lymphoma)
* Female participants who are not of child-bearing potential and female participants of child-bearing potential who have a negative serum pregnancy test within 3 days prior to initial trial treatment. Female participants of child-bearing potential and all male partners, and male participants must consent to use a medically acceptable method of contraception throughout the study period and for a minimum of 1 year after the last dose of rituximab and for a minimum of 4 months after the last dose of umbralisib.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who require immediate cytoreduction per the treating investigator.
* For patients with H. pylori related gastric extranodal marginal zone lymphoma in the absence of t(11;18): Patient must have relapsed or refractory marginal zone lymphoma despite appropriate H. pylori eradication.
* For patients with hepatitis C virus related marginal zone lymphoma: Patient must have relapsed or refractory marginal zone lymphoma despite appropriate treatment of hepatitis C virus infection.
* Active systemic therapy for another malignancy within 2 years. Local/regional therapy with curative intent such as surgical resection or localized radiation is allowed if patient is deemed at low risk for recurrence by treating physician.
* Malignancy within 3 years of study enrollment except for adequately treated basal, squamous cell carcinoma or non-melanomatous skin cancer, carcinoma in situ of the cervix, superficial bladder cancer not treated with intravesical chemotherapy or BCG within 6 months, localized prostate cancer and PSA <1.0 mg/dL on 2 consecutive measurements at least 3 months apart with the most recent one being within 4 weeks of study entry.
* Corticosteroid therapy (prednisone >10 mg daily or equivalent) is not permitted within 7 days prior to study entry. Topical, or intra-articular or inhaled corticosteroids are permitted.
* Prior allogeneic stem cell transplant.
* Inflammatory bowel disease (such as Crohn's disease or ulcerative colitis)
* Malabsorption syndromes
* Irritable bowel syndrome with greater than 3 loose stools per day as a baseline.
* Known central nervous system involvement by lymphoma.
* Evidence of histological transformation to large cell lymphoma.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to umbralisib or rituximab.
* Evidence of ongoing systemic bacterial, fungal or viral infection, except localized fungal infections of skin or nails.
* Evidence of chronic active Hepatitis B (HBV, not including patients with prior hepatitis B vaccination; or positive serum Hepatitis B antibody) or chronic active Hepatitis C infection (HCV), active cytomegalovirus (CMV), or known history of HIV. If HBc antibody is positive, the patient must be evaluated for the presence of HBV DNA (by PCR). If HCV antibody is positive, the subject must be evaluated for the presence of HCV RNA by PCR. If the patient is CMV IgG or CMV IgM positive, the subject must be evaluated for the presence of CMV DNA by PCR. Patients with positive HBc antibody and negative HBV DNA via PCR are eligible, but prophylaxis with entecavir or lamivudine is recommended. Subjects who are CMV IgG or CMV IgM positive but who are CMV DNA negative by PCR are eligible, but antiviral prophylaxis should be considered per institutional protocol.
* Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:
* Symptomatic, or history of documented congestive heart failure (New York Heart Association functional classification III-IV [see Appendix: NYHA Classifications])
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, CHF, or myocardial infarction within 6 months of enrollment.
* Concomitant use of medication known to cause QT prolongation or torsades de pointes should be used with caution and at investigator discretion.
* Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), symptomatic peripheral arterial disease, angioplasty, cardiac or vascular stenting within 6 months of enrollment.
* Psychiatric illness/social situations that would limit compliance with study requirements
* Known history of drug-induced liver injury, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by stones, cirrhosis of the liver.
* Pregnant women are excluded from this study because rituximab is an agent with known potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with rituximab or umbralisib, breastfeeding should be discontinued if the mother is treated with rituximab or umbralisib. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate | 2 years
  The frequency of patients who achieve a complete response

SECONDARY OUTCOMES:
Overall Response Rate | 2 years
  The frequency of patients who achieve a complete or partial response
Progression Free Survival | 2 years
  The median progression-free survival using Kaplan-Meier method with time of registration as time origin.
Overall Survival Rate | 2 Years
  The median overall survival using Kaplan-Meier method with time of registration as time origin.
Safety and Adverse Events: frequency, severity, and timing of adverse events | 2 years
  The nature, frequency, severity, and timing of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jacob D. Soumerai, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- See also: Link to MGH Center for Lymphoma — https://www.massgeneral.org/cancer/team/lymphoma.aspx